CLINICAL TRIAL: NCT05876390
Title: Impact of Loco-regional Anesthesia Techniques on Chronic Post-surgery in Breast Oncological Surgery: a Prospective Multicenter Observational Study
Brief Title: Impact of Regional Anesthesia on Chronic Post-operative Pain
Acronym: IRACPoP
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 603-11102022
Record Dates: First submitted 2023-03-24; First posted 2023-05-25 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast surgery; oncological breast surgery; multimodal analgesia; chronic postoperative pain
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative | interventions — Mastectomy, Segmental; Analgesia; Anti-Inflammatory Agents, Non-Steroidal; Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing oncological breast surgery: * mastectomy + reconstruction
  * simple quadrantectomy
  * quadrantectomy + sentinel lymph node biopsy
  * quadrantectomy + axillary hollowing
  * bilateral interventions will also be considered
  Interventions: Procedure: Breast surgery; Drug: analgesia

INTERVENTIONS:
Procedure: Breast surgery — Breast surgery
Drug: analgesia — Multimodal analgesia
  Other Names: • loco-regional analgesia + NSAIDs, paracetamol

SUMMARY:
Approximately 55,000 cases of breast cancer are diagnosed in Italy every year and the first-line therapy for carcinoma in situ, stage I, II and IIIA is surgical removal of the tumour. The incidence of chronic pain after breast cancer surgery is confirmed around 30%. This study aims to evaluate the impact of loco-regional anesthesia techniques in the context of multimodal analgesia in the prevention of chronic pain post-oncological breast surgery

DETAILED DESCRIPTION:
Approximately 55,000 cases of breast cancer are diagnosed in Italy every year and the first-line therapy for carcinoma in situ, stage I, II and IIIA is surgical removal of the tumour. The incidence of chronic pain after breast cancer surgery is confirmed around 30%.Persistent postsurgical pain, defined in the ICD-11 as pain that develops or increases in intensity after a surgical procedure or tissue damage and persists beyond the healing process for at least 3 months after the initial event and is considered a complication of surgery.

Several pharmacological and non-pharmacological interventions have been proposed for the prevention of the development of this complication of surgical interventions, including the intraoperative use of local anesthesia techniques in the context of multimodal analgesia.

The purpose of this multicenter prospective observational study is to evaluate, through the propensity score methodology, how much the use of loco-regional anesthesia techniques can improve the outcome, in terms of the development of chronic post-surgical pain, of patients undergoing to oncological breast surgery

ELIGIBILITY:
Inclusion criteria

* Age > 18
* Oncological breast surgery:

  * simple mastectomy,
  * mastectomy + sentinel lymph node biopsy,
  * mastectomy + axillary hollowing,
  * mastectomy + reconstruction,
  * simple quadrantectomy,
  * quadrantectomy + sentinel lymph node biopsy,
  * quadrantectomy + axillary hollowing,
  * bilateral interventions will also be considered) Exclusion
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing oncological breast surgery
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic postoperative pain after major breast surgery | 6 - 12 months
  Incidence of chronic post-surgical pain after major breast surgery (definition: pain that persists at least 3 months after surgery; pain that was not present before surgery or that has different characteristics from pain before surgery or that has increased intensity than before the operation; the pain is localized in the area of the surgical site or in its radiation; other possible causes of pain are excluded)

SECONDARY OUTCOMES:
Acute post-operative pain | 2, 6, 12 and 24 hours
  Acute postoperative pain. NRS Numerical Rating Scale (0-10; 0 =better 10= worse outcome)
Chronic post-operative pain | 3,6,9,12 months) at rest and on mobilization
  Pain both at rest and on mobilization month3, month6, month9 and month12 after surgery. Numerical Rating Scale (0-10; 0 =better 10= worse outcome)
Quality of life score | Quality of recovery score (QoR 15)
  Quality of recovery score-15 (QoR 15; scale 0-150; 0=better 150=worse outcome)
Remifentanyl | Intraoperative
  Intraoperative use of remifentanil. Intraoperative quantitative use of remifentanyl (total micrograms; the lesser the better)
Opioid | hour2, hour 6, hour 12 and hour 24 after surgery
  Postoperative opioid use. (opioid oral morphine milligram equivalent (MME); the lesser the better)

CONTACTS AND LOCATIONS:
Locations (1):
- ASST GOM Niguarda, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Yes
The results obtained will be used for a scientific publication and for the elaboration of a specialist degree thesis in Anesthesia and Intensive Care
Supporting Information: Study Protocol, SAP